CLINICAL TRIAL: NCT01559662
Title: A Prospective Randomized Controlled Trial of Sugared Chewing Gum on Gastrointestinal Recovery After Major Colorectal Surgery in Patients Managed With Early Enteral Feeding
Brief Title: Effect of Sugared Chewing Gum on Gastrointestinal Recovery After Major Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Pricipal investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMCGumStudy
Record Dates: First submitted 2012-03-16; First posted 2012-03-21 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Ileus
Keywords: chewing gum; ileus; gastrointestinal function; colorectal surgery; abdominal surgery
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugared Chewing Gum (Experimental): Patient asked to chew sugared chewing gum postoperative day 1 to 7, 3 times a day, 45 minutes at a time
  Interventions: Dietary Supplement: Sugared Chewing Gum (Juicy Fruit)
- No Gum (No Intervention): No gum given, routine postoperative care provided

INTERVENTIONS:
Dietary Supplement: Sugared Chewing Gum (Juicy Fruit) — One stick of gum, 3 times daily from Postoperative day 1 to 7
  Arms: Sugared Chewing Gum

SUMMARY:
The Purpose of this study is to evaluate the effect of gum chewing on recovery of gastrointestinal function in patient undergoing major colorectal surgery. The investigators hypothesize that patients who chew gum after major colorectal surgery will have faster recovery of gastrointestinal function.

ELIGIBILITY:
Inclusion Criteria:

* Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form
* American Society of Anesthesiologists (ASA) Class I-III (Appendix III);
* Due to undergo small and/or large partial bowel resection via laparotomy or laparoscopy

Exclusion Criteria:

* Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures
* American Society of Anesthesiologists (ASA) Class IV or V;
* History of abdominal carcinomatosis
* History of radiation enteritis
* Children < 18 or adults > 85 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time (in hours) to tolerating a low residue diet | 30 day postoperative period
  Time measured from end of operation to patient tolerating 50% of a low residue diet without emesis in 24 hours

SECONDARY OUTCOMES:
Time (in hours) to passage of flatus | 30 day postoperative period
  Time from end of operation to first passage of flatus (reported by patient)
Time (hours) to first bowel movement | 30 day postoperative period
  Time (hours) from end of operation to first bowel movement
Daily Appetite Assessment | Postoperative day 1 - 7
  Patient asked to record appetite on a scale from 0 (no appetite) to 10 (appetite as good as can be)
Daily pain assessment | Postoperative day 1 - 7
  Patient asked to rate pain on VAS scale from 0 (no pain) to 10 (pain as bad as can be)
Daily nausea assessment | Postoperative day 1 - 7
  Patient asked to rate nausea on a scale from 0 (no nausea) to 10 (nausea as bad as can be)
Major or Minor Medical and Surgical Complications | 30 day postoperative period
Length of postoperative hospitalization in days | Duration of postoperative hospitalization (expected average of 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States